CLINICAL TRIAL: NCT04912349
Title: Comparison of Transurethral Split of the Prostate Versus Transurethral Resection of the Prostate for Treatment of Benign Prostatic Hyperplasia in a Small Prostate Volume: A Prospective Controlled Study
Brief Title: Comparison of TUSP Versus TURP for Treatment of Benign Prostatic Hyperplasia in a Small Prostate Volume
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-525
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Patients received the transurethral split of the prostate(TUSP) treatment.
  Interventions: Procedure: TUSP
- Control Group (Active Comparator): Patients received the transurethral resection of the prostate(TURP) treatment.
  Interventions: Procedure: TURP

INTERVENTIONS:
Procedure: TUSP — Patients received the transurethral split of the prostate(TUSP) treatment.
  Arms: Test Group
Procedure: TURP — Patients received the transurethral resection of the prostate(TURP) treatment.
  Arms: Control Group

SUMMARY:
Comparison of transurethral split of the prostate versus transurethral resection of the prostate for treatment of benign prostatic hyperplasia in a small prostate volume: A prospective controlled study

DETAILED DESCRIPTION:
Transurethral resection of the prostate (TURP) was considered as the golden standard to treat benign prostatic hyperplasia (BPH) for decades. However, TURP was associated with low efficiency to alleviate the lower urinary tract symptoms and a significantly higher risk of bladder neck contracture (BNC) for patients with small-volume BPH. We aimed to compare the therapeutic effect of transurethral split of the prostate (TUSP) with TURP for patients with small-volume BPH (<30 ml).

In this study, some selected small-volume BPH patients were randomly divided into two groups (TUSP and TURP group). The patient's baseline characteristics and perioperative outcomes were recorded. The follow-up was made at 6 months, 1 year and 2 years after surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Benign prostatic hyperplasia patients with surgical indication
* Maximum flow rate <12ml/s
* Prostate volume <30ml
* The international prostate symptoms score>21
* Medication of α-adrenergic blockers for at least 3 months

Exclusion Criteria:

* Acute prostatitis and urethritis
* Neurogenic bladder
* Abnormal prostate-specific antigen level
* Urethral injury history

Ages: 35 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
international prostate symptoms score（IPSS） | within 24 months after surgery
  Measuring the International Prostate Symptoms Score by a questionnaire (which minimum value is zero and the maximum value is 35; higher scores mean a worse outcome)
maximum urinary flow rate（Qmax） | within 24 months after surgery
  Measuring the maximum urinary flow rate by a urodynamic study

CONTACTS AND LOCATIONS:
Overall Officials: Jiaming Wen, Dr., Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No